CLINICAL TRIAL: NCT04631705
Title: A Phase 1/2a Trial of the Inhaled Administration of the SARS-CoV-2-Neutralizing Monoclonal Antibody DZIF-10c in SARS-CoV-2-Infected and -Uninfected Individuals
Brief Title: SARS-CoV-2-Neutralizing Monoclonal COVID-19 Antibody DZIF-10c by Inhalation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Change in viral variant epidemiology
Sponsor: University of Cologne (Other)
Collaborators: ZKS Köln (Other); Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Florian Klein, Investigator, University of Cologne
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: Uni-Koeln-4370
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-06

CONDITIONS: SARS-CoV-2 Infection
Keywords: SARS-CoV-2; Covid-19; Monoclonal Antibody; Inhalation
MeSH Terms: conditions — COVID-19; Respiratory Aspiration | interventions — BI 767551

STUDY DESIGN:
Intervention Model Description: This study consists of an open-label dose escalation phase in both healthy volunteers (Groups 1A-1C) and SARS-CoV-2-infected participants (Groups 2A-2C).
  After completion of the dose escalation phase, SARS-CoV-2-infected individuals will be enrolled into a randomized placebo-controlled expansion cohort (Group 2D).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1A (uninfected) - low dose (Experimental): SARS-CoV-2-uninfected volunteers will receive a single dose of DZIF-10c by inhalation
  Interventions: Biological: DZIF-10c
- Group 1B (uninfected) - mid dose (Experimental): SARS-CoV-2-uninfected volunteers will receive a single dose of DZIF-10c by inhalation
  Interventions: Biological: DZIF-10c
- Group 1C (uninfected) - high dose (Experimental): SARS-CoV-2-uninfected volunteers will receive a single dose of DZIF-10c by inhalation
  Interventions: Biological: DZIF-10c
- Group 2A (infected) - low dose (Experimental): SARS-CoV-2-infected volunteers will receive a single dose of DZIF-10c by inhalation
  Interventions: Biological: DZIF-10c
- Group 2B (infected) - mid dose (Experimental): SARS-CoV-2-infected volunteers will receive a single dose of DZIF-10c by inhalation
  Interventions: Biological: DZIF-10c
- Group 2C (infected) - high dose (Experimental): SARS-CoV-2-infected volunteers will receive a single dose of DZIF-10c by inhalation
  Interventions: Biological: DZIF-10c
- Group 2D (infected) (Experimental): SARS-CoV-2-infected volunteers will be randomized 1:1:1 to receive DZIF-10c by inhalation and infusion, DZIF-10c by inhalation and placebo by infusion, or placebo by inhalation and infusion
  Interventions: Biological: DZIF-10c; Drug: Placebo

INTERVENTIONS:
Biological: DZIF-10c — Inhaled administration of the human monoclonal antibody DZIF-10c
Biological: DZIF-10c — Intravenous administration of the human monoclonal antibody DZIF-10c
  Arms: Group 2D (infected)
Drug: Placebo — Inhalation of DZIF-10c diluent as placebo
  Arms: Group 2D (infected)
Drug: Placebo — Intravenous infusion of sterile normal saline (NaCl 0.9%) as placebo
  Arms: Group 2D (infected)

SUMMARY:
This is the first-in-human phase 1/2a trial of the inhaled administration of the SARS-CoV-2-neutralizing monoclonal antibody DZIF-10c in healthy volunteers and SARS-CoV-2-infected individuals. It will evaluate the safety, pharmacokinetic profile, immunogenicity, and antiviral activity of DZIF-10c.

DETAILED DESCRIPTION:
The phase 1 component of this trial consists of a single-inhalation open-label dose-escalation phase (Groups 1A-1C and Groups 2A-2C). Subsequently, the highest tolerated dose tested will be administered to an expansion cohort of SARS-CoV-2-infected individuals (Group 2D). In this randomized and blinded group, participants will receive DZIF-10c or placebo both by inhalation and intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

Groups 1A-1C

* Age 18-65.
* SARS-CoV-2-RNA negative naso- or oropharyngeal swab obtained within 3 calendar days before study drug administration by NAAT (e.g., qRT-PCR).
* Non-reactivity of serum antibodies (IgG; and IgA and/or IgM when tested) against SARS-CoV-2 by serological assay at screening.

Groups 2A-2D

* Age 18-70.
* SARS-CoV-2-RNA positive naso- or oropharyngeal swab obtained within 3 calendar days before study drug administration by NAAT (e.g., qRT-PCR).
* Onset of COVID-19 symptoms (e.g., sore throat, cough, fever, chills, fatigue, dys- or anosmia, dys- or ageusia, headache, muscle pain, gastrointestinal symptoms) within 7 days prior to study drug administration or Non-reactivity of serum or plasma antibodies (IgG; and IgA and/or IgM when tested) against SARS-CoV-2 by serological assay at screening.
* Disease severity score 1-4 as defined by the WHO Clinical Progression Scale (WHO, Lancet Inf Dis 2020)

Exclusion Criteria (all groups):

* Known hypersensitivity to any constituent of the investigational medicinal product.
* Hepatitis B infection indicated by detectable HBsAg (Hepatitis B surface antigen) in blood.
* Detectable antibodies against hepatitis C virus in blood unless active hepatitis C is ruled out by negative HCV-RNA.
* HIV infection indicated by detectable HIV antigen and/or HIV antibodies in blood.
* Neutrophil count ≤1,000 cells/µl
* Hemoglobin ≤10 g/dl
* Platelet count ≤100,000 cells/µl
* ALT ≥2.0 x ULN
* AST ≥2.0 x ULN
* Total bilirubin ≥1.5 ULN
* eGFR <60 ml/min/1.73m2
* Pregnancy or lactation.
* Any vaccination within 14 days prior to DZIF-10c administration.
* Receipt of any SARS-CoV-2 vaccine or SARS-CoV-2 monoclonal antibody in the past.
* Diagnosis of bronchial asthma or history of bronchial hyperresponsiveness, COPD, pulmonary fibrosis, or other chronic lung diseases.
* Any chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer.
* History of systemic corticosteroids, immunosuppressive anti-cancer, or other medications considered significant by the trial physician within the last 6 months (a single administration of systemic corticosteroids within ≤6 months and ≥4 weeks of enrollment is acceptable).
* Participation in another clinical trial of an investigational medicinal product within the past 12 weeks or expected participation during this study.
* Dependency on the principal investigator or study staff; or site personnel directly affiliated with this trial.
* Legally incapacitated individuals
* Individuals held in an institution by legal or official order
* If engaging in sexual activity that could result in pregnancy, inability or unwillingness to comply with the requirements for highly effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Fätkenheuer, MD, Principal Investigator — University of Cologne
Locations (6):
- Germany (6):
  - University Hospital Gießen and Marburg, Giessen, Hesse
  - University Hospital Cologne, Cologne, North Rhine-Westphalia
  - University Hospital Düsseldorf, Düsseldorf
  - University Hospital Frankfurt, Frankfurt am Main
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - LMU Munich University Hospital, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kreer C, Zehner M, Weber T, Ercanoglu MS, Gieselmann L, Rohde C, Halwe S, Korenkov M, Schommers P, Vanshylla K, Di Cristanziano V, Janicki H, Brinker R, Ashurov A, Krahling V, Kupke A, Cohen-Dvashi H, Koch M, Eckert JM, Lederer S, Pfeifer N, Wolf T, Vehreschild MJGT, Wendtner C, Diskin R, Gruell H, Becker S, Klein F. Longitudinal Isolation of Potent Near-Germline SARS-CoV-2-Neutralizing Antibodies from COVID-19 Patients. Cell. 2020 Sep 17;182(6):1663-1673. doi: 10.1016/j.cell.2020.08.046. No abstract available. PMID 32946786
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- 1A: Healthy, 50 mg Inh.; 1B: Healthy, 100 mg Inh.; 1C: Healthy, 250 mg Inh.: Open label, SARS-CoV-2 negative, DZIF-10c dose administered by inhalation
- 2A: Infected, 50 mg Inh.; 2B: Infected, 100 mg Inh.; 2C: Infected, 250 mg Inh.: Open label, SARS-CoV-2-infected, DZIF-10c dose administered by inhalation
- 2D: Infected, Placebo Inh., Placebo i.v.: Double blind and randomized, SARS-CoV-2-infected, placebo by inhalation, placebo by i.v. infusion
- 2D: Infected, 250 mg Inh., Placebo i.v.: Double blind and randomized, SARS-CoV-2-infected, DZIF-10c by inhalation, placebo by i.v. infusion
- 2D: Infected, 250 mg Inh., 40 mg/kg i.v.: Double blind and randomized, SARS-CoV-2-infected, DZIF-10c by inhalation, DZIF-10c by i.v. infusion
Period: Overall Study
Arm/Group | 1A: Healthy, 50 mg Inh. | 1B: Healthy, 100 mg Inh. | 1C: Healthy, 250 mg Inh. | 2A: Infected, 50 mg Inh. | 2B: Infected, 100 mg Inh. | 2C: Infected, 250 mg Inh. | 2D: Infected, Placebo Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v.
Started | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 8 | 9
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 9 | 8 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1A: Healthy, 50 mg Inh. | 1B: Healthy, 100 mg Inh. | 1C: Healthy, 250 mg Inh. | 2A: Infected, 50 mg Inh. | 2B: Infected, 100 mg Inh. | 2C: Infected, 250 mg Inh. | 2D: Infected, Placebo Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v. | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 8 | 9 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 43 [29 to 44] | 33 [32 to 44] | 27 [20 to 29] | 35 [30 to 62] | 39 [25 to 42] | 41 [32 to 46] | 34 [28 to 36] | 32 [29 to 46] | 28 [27 to 38] | 33 [28 to 42.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 2 | 4 | 15
  Male | 3 | 2 | 1 | 2 | 1 | 2 | 8 | 6 | 5 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 8 | 9 | 45

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Any AE Within 7 d of Study Drug Administration
Time Frame: Over first 7 days after study drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Healthy, 50 mg Inh. | 1B: Healthy, 100 mg Inh. | 1C: Healthy, 250 mg Inh. | 2A: Infected, 50 mg Inh. | 2B: Infected, 100 mg Inh. | 2C: Infected, 250 mg Inh. | 2D: Infected, Placebo Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v.
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 10 | 8 | 9
Participants | 2 | 1 | 1 | 3 | 1 | 0 | 6 | 3 | 3

2. Secondary Outcome: DZIF-10c Area Under the Curve
Description: Area under the Curve based on serum antibody levels; 4 hour post dose collected in groups 1A-1C and 2A-2C, 1 hour post dose in group 2D (timings referring to last adminstered product); 21 day post dose only in groups 1A-1C. Geometric mean values were only calculated for groups in which at least three individuals with detectable serum levels were included.
Time Frame: 0, 1, and 4 hours post dose; 1, 3, 7, 14, 21, 28, 56, 90 days post dose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/ml
Arm/Group | 1A: Healthy, 50 mg Inh. | 1B: Healthy, 100 mg Inh. | 1C: Healthy, 250 mg Inh. | 2A: Infected, 50 mg Inh. | 2B: Infected, 100 mg Inh. | 2C: Infected, 250 mg Inh. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v.
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 9
μg*h/ml | NA (NA) — Data could not be calculated because DZIF-10c in serum was only detected in a single individual and only at two time points (day 3 and day 7 post dose). | NA (NA) — Data could not be calculated because DZIF-10c in serum was only detected in a single individual who also had reactivity in the test determined to measure DZIF-10c serum levels prior to DZIF-10c administration (i.e., background reactivity that prevented accurate determination of DZIF-10c levels). | 284 (18.2) | NA (NA) — Data could not be calculated because DZIF-10c was not detected in serum in any of the participants. | 199 (NA) — Data calculated from single participant - therefore no coefficient of variation can be determined. No DZIF-10c in serum could be detected in the remaining two participants. | NA (NA) — Data available from only two participants, therefore no geometric mean and coefficients of variation calculated. Individual values for AUC were 220 and 319 μg*h/ml. DZIF-10c could not be detected in serum in the remaining individual. | 225 (39.2) | 174000 (14.5)

3. Secondary Outcome: Anti-Drug Antibody Development
Description: Individuals developing anti-drug antibodies
Time Frame: 0, 14, 28, 56, 90 days post dose
Measure: Count of Participants; unit: Participants
Arm/Group | 1A: Healthy, 50 mg Inh. | 1B: Healthy, 100 mg Inh. | 1C: Healthy, 250 mg Inh. | 2A: Infected, 50 mg Inh. | 2B: Infected, 100 mg Inh. | 2C: Infected, 250 mg Inh. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v.
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 8 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Time-weighted SARS-CoV-2 Viral Load Change From Baseline
Description: Time-weighted change of SARS-CoV-2 viral load from baseline in nasopharyngeal swab samples as determined by the SARS-CoV-2 E gene; based on a parametric analysis of covariance model with corresponding baseline viral load, antibody status at baseline, and treatment; determined as the adjusted mean area over the curve (AOC) for samples collected at baseline and 1, 3, 7, 14, 28 days post dose
Time Frame: 0, 1, 3, 7, 14, 28 days post dose
Measure: Mean (Standard Error); unit: log10 cp/ml
Arm/Group | 2D: Infected, Placebo Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v.
Number analyzed (Participants) | 10 | 8 | 9
log10 cp/ml
  Over 7 days | -1.932 (0.263) | -2.100 (0.294) | -1.716 (0.268)
  Over 14 days | -2.780 (0.238) | -3.044 (0.267) | -2.786 (0.244)
  Over 28 days | -3.616 (0.126) | -3.652 (0.142) | -3.652 (0.129)

5. Secondary Outcome: MMRM SARS-CoV-2 Viral Load Change From Baseline
Description: Change of SARS-CoV-2 viral load from baseline in nasopharyngeal swab samples as determined by the SARS-CoV-2 E gene; based on Mixed Model for Repeated Measures (MMRM) with fixed effects for antibody status at BL, LOG10 (viral load) at BL and interaction with visit, treatment-by-visit interaction, and random effect for patient; samples collected at baseline and 1, 3, 7, 14, 28 days post dose
Time Frame: 0, 1, 3, 7, 14, 28 days post dose
Measure: Mean (Standard Error); unit: Adjusted log10 VL (cp/ml)
Arm/Group | 2D: Infected, Placebo Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v.
Number analyzed (Participants) | 10 | 8 | 9
Adjusted log10 VL (cp/ml)
  Over 7 days | -3.4 (0.4) | -3.4 (0.5) | -3.2 (0.5)
  Over 14 days | -4.4 (0.1) | -4.1 (0.1) | -4.4 (0.1)
  Over 28 days | -4.4 (0.3) | -4.3 (0.3) | -4.4 (0.3)

ADVERSE EVENTS:
Time Frame: 90 days (treatment-emergent adverse events: All adverse events after drug intake until final study visit)
Description: Participants were queried about potential Adverse Events at all study visits.
Arm/Group | 1A: Healthy, 50 mg Inh. | 1B: Healthy, 100 mg Inh. | 1C: Healthy, 250 mg Inh. | 2A: Infected, 50 mg Inh. | 2B: Infected, 100 mg Inh. | 2C: Infected, 250 mg Inh. | 2D: Infected, Placebo Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., Placebo i.v. | 2D: Infected, 250 mg Inh., 40 mg/kg i.v.
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/10 | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/10 | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 2/3 | 3/3 | 2/3 | 2/3 | 7/10 | 5/8 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1A: Healthy, 50 mg Inh. (N=3) | 1B: Healthy, 100 mg Inh. (N=3) | 1C: Healthy, 250 mg Inh. (N=3) | 2A: Infected, 50 mg Inh. (N=3) | 2B: Infected, 100 mg Inh. (N=3) | 2C: Infected, 250 mg Inh. (N=3) | 2D: Infected, Placebo Inh., Placebo i.v. (N=10) | 2D: Infected, 250 mg Inh., Placebo i.v. (N=8) | 2D: Infected, 250 mg Inh., 40 mg/kg i.v. (N=9)
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Inflammation (General disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 2 (2) | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (3) | 0 | 2 (2)
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Aphasia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 (2) | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (3) | 0 | 0 | 2 (2) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0 | 0 | 5 (6) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (3) | 0
Headache (Nervous system disorders) | 1 (1) | 0 | 0 | 2 (2) | 0 | 1 (1) | 2 (3) | 2 (2) | 3 (6)
Sciatica (Nervous system disorders) | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 (2) | 0 | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1)
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0
Gonococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 (1) | 0 | 0

LIMITATIONS AND CAVEATS:
- Small sample size, further reduced by early termination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications by PIs are to be submitted to the sponsor for review at least 30 days prior to planned disclosure. Modifications suggested by the sponsor should be considered unless they affect the scientific character or neutrality of the publication. A maximum embargo period of 90 days is applicable only if disclosure would affect (potential) intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT04631705/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT04631705/SAP_001.pdf